CLINICAL TRIAL: NCT05816785
Title: A Pilot Window of Opportunity Study of Imatinib in Combination With Cetuximab in Patients With Squamous Cell Carcinomas of the Head and Neck
Brief Title: Pilot Study of Imatinib Cetuximab Combo for H & N Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-1590; 1R01CA262292-01A1 (NIH); NCI-2023-01888 (Registry Identifier: CTRP); UW22118 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); Protocol Version 7/2/2025 (Other: UW Madison)
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Imatinib Mesylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imatinib Cetuximab Combination (Experimental): Participants will receive two doses of CTX and a minimum of an 8 day (maximum 14 day) course of imatinib prior to definitive surgery or definitive radiation/chemoradiation.
  Interventions: Drug: Cetuximab; Drug: Imatinib

INTERVENTIONS:
Drug: Cetuximab — Week 1: loading dose of 400mg/m2; Week 2: 250mg/m2
Drug: Imatinib — 400 mg orally daily

SUMMARY:
The goal of this clinical trial is to find if levels of a protein called AXL in tumor cells relate to how tumors respond to cetuximab (CTX) combined with imatinib in participants with head and neck cancer. This interventional study will occur in the time between diagnosis of your cancer and surgery to remove your tumor or radiation or chemoradiation treatment of your primary cancer.

Participants will undergo a research blood draw and a research biopsy as part of the screening process, and will be in this research study for approximately 13 to 16 months.

DETAILED DESCRIPTION:
This is a 'window of opportunity' pilot study of oral imatinib (400 mg per day) plus cetuximab (CTX) (400mg/m2 loading dose [dose 1] and 250mg/m2 [dose 2]) for patients with head and neck squamous cell carcinoma (HNSCC) undergoing definitive surgery or radiation for treatment of their cancer. The primary objective is to determine the proportion of patients with a response to imatinib plus CTX in pre-treatment and post-treatment samples obtained as part of a window of opportunity clinical study in head and neck cancer (HNC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years at the time of consent.
* Histological confirmation of squamous cell carcinoma of the head and neck.

  * For those patients with oropharyngeal cancer, subjects must have either
  * HPV-negative status by p16 expression or HPV-DNA Expression.
  * HPV-positive status by p16 expression AND a >10 pack year smoking history.
* Subjects must be appropriate candidates for definitive curative intent treatment, either via surgical resection, definitive radiation therapy alone, or definitive concurrent chemoradiation therapy.
* For the screening research biopsy, subjects must have sufficient tumor volume (approximately 10 cc) to accommodate at minimum 2-3 core samples for the research biopsy.
* For the post-treatment (CTX/Imatinib) research biopsy, subjects who are scheduled to receive definitive radiation therapy (+/- concurrent chemotherapy) are required to have sufficient tumor volume to accommodate at minimum 2-3 core samples for the research biopsy.
* Demonstrate adequate organ function; all screening labs to be obtained within 28 days prior to registration.

Exclusion Criteria:

* Subjects with a diagnosis of nasopharyngeal carcinoma, advanced cutaneous squamous cell carcinoma of the head and neck, or salivary gland tumors are excluded from this study.
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol.
* Prior chemotherapy, radiotherapy, or major surgery within 8 weeks of study enrollment or those who have not recovered (to grade ≤ 1 or baseline) from clinically significant adverse events due to agents administered more than 8 weeks earlier (alopecia and fatigue excluded). Clinical significance to be determined by the study investigator.
* Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Subjects who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imatinib or CTX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Ki67 from pre- versus post-imatinib/cetuximab treated tumors | 6 months after last research biopsy
  The change in Ki67 is calculated as the ratio of pre- to post- treatment Ki67 index

SECONDARY OUTCOMES:
Adverse Events that are probably related to CTX and imatinib prior to the start of definitive concurrent chemoradiation therapy or surgical resection | Through study completion, an average of 2 years
  Count of adverse events that are probably related to the regimen
Rate of hospital re-admissions | Up to 28 days after surgery
  For subjects undergoing definitive surgical resection, rate of hospital re-admissions for wound care or surgical complications attributed to imatinib plus cetuximab (such as fistula or deep cellulitis) within 28 days after surgery
Objective response rate (ORR) | Diagnosis, 48 hours prior to surgery or radiation
  Measured by clinical examination
Objective response rate (ORR) | Diagnosis, 48 hours prior to surgery or radiation
  Measured by clinical measurements

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes